CLINICAL TRIAL: NCT03059251
Title: An Observational Study of the Safety and Effectiveness of Obinutuzumab in Patients With Chronic Lymphocytic Leukemia Treated in Argentina
Brief Title: Observational Study: Safety and Effectiveness of Obinutuzumab in Chronic Lymphocytic Leukemia in Argentina
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30187
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL, obinutuzumab, treatment
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Obinutuzumab: All participants with chronic lymphocytic leukemia (CLL) who have received the indication for treatment with Obinutuzumab, as per routine clinical practice in Argentina.
  Interventions: Biological: Obinutuzumab

INTERVENTIONS:
Biological: Obinutuzumab — Obinutuzumab will be administered as intravenous infusion for 6 cycles (28 days per cycle): 100 milligrams (mg) on day 1 Cycle 1, 900 mg on day 2 Cycle 1, 1000 mg on days 8 and 15 of Cycle 1, and 1000 mg on day 1 of Cycles 2-6.
  Other Names: Gazyva®

SUMMARY:
This observational study aims to study the effectiveness and safety of Obinutuzumab in common clinical practice settings in Argentina. The study population comprises all patients with chronic lymphocytic leukemia (CLL) that have received the indication for treatment with Obinutuzumab as per routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Have received at least one dose of Obinutuzumab as per local label and clinical practice.

Exclusion Criteria:

* Included in clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic lymphocytic leukemia (CLL) who have received the indication for treatment with Obinutuzumab as per routine clinical practice in Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 2 months after completion of 6 treatment cycles (up to approximately 8 months)
  Overall response rate was defined as percentage of participants with complete response (CR) or partial response (PR). CR was defined as peripheral blood lymphocytes below 4 x 10^9/liter (L), absence of significant lymphadenopathy, no hepatomegaly, no splenomegaly, absence of disease or B symptoms, neutrophils >1.5 x 10^9/L, platelets >100 x 10^9/L, hemoglobin >11 grams/deciliter (g/dl) and bone marrow at least normocellular for age. PR was defined as >=50% decrease in peripheral blood lymphocyte count, >/=50% reduction in lymphadenopathy, >/=50% reduction of liver enlargement and/or >/=50% reduction of spleen enlargement, plus at least one of the following: neutrophils >1.5 x 10^9/L or >/=50% increase, or platelets >100 x 10^9/L or ≥50% increase, or hemoglobin 11 g/dl or >/=50% increase. Overall response rate = CR + PR
Percentage of Participants With Adverse Events (AEs) | Up to 24 months
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

SECONDARY OUTCOMES:
Complete Response Rate | Up to 2 months after completion of 6 treatment cycles (up to approximately 8 months)
  CR was defined as peripheral blood lymphocytes below 4 x 10^9/liter (L), absence of significant lymphadenopathy, no hepatomegaly, no splenomegaly, absence of disease or B symptoms, neutrophils >1.5 x 10^9/L, platelets >100 x 10^9/L, hemoglobin 11 g/dl and bone marrow at least normocellular for age.
Partial Response Rate | Up to 2 months after completion of 6 treatment cycles (up to approximately 8 months)
  PR was defined as >=50% decrease in peripheral blood lymphocyte count from the pre-treatment value, >/=50% reduction in lymphadenopathy, >/=50% reduction of liver enlargement and/or >/=50% reduction of spleen enlargement, plus at least one of the following: neutrophils >1.5 x 10^9/L or >/=50% increase, or platelets >100 x 10^9/L or ≥50% increase, or hemoglobin 11 g/dl or >/=50% increase.
Progression-free Survival (PFS) | After the completion of treatment, at 12 and 24 months after start of treatment
  PFS is defined as the time from the first dose of treatment to the first occurrence of progression, or death from any cause as assessed by the physician. Progressive disease is defined by any of the following: >/=50% increase in the absolute number of lymphocytes, appearance of new palpable lymph nodes (>15 mm in longest diameter) or any new extra nodal lesion, >/=50% increase in the longest diameter of any previous site of clinically significant lymphadenopathy, >/=50% increase in the enlargement of the liver and/or spleen, transformation to a more aggressive histology, after treatment, the progression of any cytopenia (a decrease of hemoglobin levels >2 g/dL or <10 g/dL or a decrease of platelet counts >50% or <100 x 10x9/L or by a decrease of neutrophil counts >50% or <1.0 x 10^9/L), excluding immune causes.
Median Duration of Response | Up to 24 months
  Duration of response is defined as the time from the date the response (either CR or PR) was first recorded until the date of disease progression or death due to any cause. Disease progression is defined by any of the following: >/=50% increase in the absolute number of lymphocytes, appearance of new palpable lymph nodes (>15 mm in longest diameter) or any new extra nodal lesion, >/=50% increase in the longest diameter of any previous site of clinically significant lymphadenopathy, >/=50% increase in the enlargement of the liver and/or spleen, transformation to a more aggressive histology, after treatment, the progression of any cytopenia (a decrease of hemoglobin levels >2 g/dL or <10 g/dL or a decrease of platelet counts >50% or <100 x 10x9/L or by a decrease of neutrophil counts >50% or <1.0 x 10^9/L), excluding immune causes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Argentina (3):
  - Clínica Peuyrredón, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Municipal Teodoro Alvarez, Buenos Aires